CLINICAL TRIAL: NCT00658541
Title: A Randomized, Two-way Crossover, Single-dose, Open-label Study to Evaluate the Relative Bioequivalence of a Test Tablet Formulation of Zolpidem Tartrate 10mg, Compared to an Equivalent Dose of Ambien® in Fed, Healthy, Adult Subjects
Brief Title: Fed Bioequivalence Study of Zolpidem Tartrate Tablets and Ambien® Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 04065
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2010-01-20 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Healthy; Therapeutic Equivalency
MeSH Terms: interventions — Zolpidem; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem Tartrate 10 mg Tablets (Experimental): A single dose of zolpidem tartrate 10 mg administered following an overnight fast of at least 10 hours and a standardized, high fat breakfast.
  Interventions: Drug: Zolpidem Tartrate 10 mg tablet
- Zolpidem Tartrate (Ambien®) 10 mg Tablets (Active Comparator): A single dose of Ambien® 10 mg administered following an overnight fast of at least 10 hours and a standardized, high fat breakfast.
  Interventions: Drug: Zolpidem Tartrate 10 mg tablet (Ambien®)

INTERVENTIONS:
Drug: Zolpidem Tartrate 10 mg tablet — 10 mg tablet administered following an overnight fast of at least 10 hours and a standardized, high fat breakfast.
  Arms: Zolpidem Tartrate 10 mg Tablets
Drug: Zolpidem Tartrate 10 mg tablet (Ambien®) — 10 mg tablet administered following an overnight fast of at least 10 hours and a standardized, high fat breakfast.
  Other Names: Ambien®
  Arms: Zolpidem Tartrate (Ambien®) 10 mg Tablets

SUMMARY:
The purpose of this study is to compare the bioequivalence of a test formulation of zolpidem tartrate tablets to an equivalent oral dose of the commercially available Ambien® (zolpidem tartrate tablets)in adult subjects under fed conditions.

DETAILED DESCRIPTION:
The purpose of this study is to compare the bioequivalence of a test formulation of zolpidem tartrate tablets to an equivalent oral dose of the commercially available Ambien® (zolpidem tartrate tablets)in adult subjects under fed conditions.

Thirty-eight healthy, non-smoking, non-obese male and female volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two zolpidem tartrate dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, following an overnight fast of at least 10 hours and a standardized, high fat breakfast, subjects will receive either a single oral dose of the test formulation, zolpidem tartrate (1 x 10 mg tablet) or a single oral dose of the reference formulation, Ambien® (1 x 10 mg tablet). After a 7 day washout period, on the morning of Day 8 following an overnight fast of at least 10 hours and a standardized, high fat breakfast, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 12 hours post dose at times sufficient to adequately define the pharmacokinetics of zolpidem tartrate. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drugs and/or procedures. Blood pressure and pulse rate will be obtained prior to dosing and at 0.5, 1, 2, 4 and 12 hours post-dose. All adverse events whether elicited by query, spontaneously reported or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or Female; similar proportions of each preferred
* Age: At least 18 years
* Weight: must be 15% of ideal weight for height and frame
* Subjects must be in good health and physical condition as determined by medical history
* Subjects must read and sign the Consent Form

Exclusion Criteria:

* history of treatment for alcoholism, substance abuse, or drug abuse within past 24 months
* history of malignancy, stroke, diabetes, cardiac, renal or liver disease
* history of GERD, malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease
* history of treatment for asthma within the past five (5) years
* history of mental depression, pulmonary disease, sleep apnea
* females who are pregnant or lactating
* history of hypersensitivity to zolpidem tartrate, or any hypnotic or sedative
* conditions upon screening which might contraindicate or require that caution be used in the administration of zolpidem tartrate, including sitting systolic blood pressure below 90 mm Hg, or diastolic pressure below 50 mm Hg; heart rate less than 50 beats per minute after a 5-minute rest in a seated position
* inability to read and/or sign the consent form
* treatment with any other investigation drug during the four (4) weeks prior to the initial dosing for this study
* subjects who have donated blood within four (4) weeks prior to the initial dosing for this study
* subjects who smoke or use tobacco products or are currently using nicotine products (patches, gums, etc.) Three (3) months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-05; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets: On the morning of Day 1 following an an overnight fast of at least 10 hours and a standardized, high-fat breakfast, each subject received one tablet of the test formulation, zolpidem tartrate 10 mg, followed by a 7 day washout period. Then, on the morning of Day 8 following an overnight fast of at least 10 hours and a standardized, high-fat breakfast, each subject received a single tablet of the reference formulation, Ambien® 10 mg.
- Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets: On the morning of Day 1 following an overnight fast of at least 10 hours and a standardized, high fat breakfast, each subject received one tablet of the reference formulation, Ambien® 10 mg, followed by a 7 day washout period. Then, on the morning of Day 8 following an overnight fast of at least 10 hours and a standardized, high fat breakfast, each subject received a single tablet of the test formulation, zolpidem tartrate 10 mg.
Period: First Intervention
Arm/Group | Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets | Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets | Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets
Started | 19 | 19
Completed | 18 | 17
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets | Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zolpidem Tartrate 10 mg Tablets and Ambien® 10 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either zolpidem tartrate 10 mg or Ambien® 10 mg following an overnight fast of at least 10 hours and a standardized, high fat breakfast.
Arm/Group | Zolpidem Tartrate 10 mg Tablets and Ambien® 10 mg Tablets
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.21 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Zolpidem Tartrate
Description: The maximum or peak concentration that zolpidem tartrate reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing (hour 0), and then at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 4, 5, 6, 8, 10, and 12 hours after dose administration
Population: Plasma concentration data for 35 of 38 participants were used in the statistical analysis. One subject dropped from the study during Period I and two subjects dropped from the study after Period I.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Zolpidem Tartrate 10 mg Tablets: Each subject received one tablet of zolpidem tartrate 10 mg after an overnight fast of at least 10 hours and a standardized, high fast breakfast.
- Ambien® 10 mg Tablets: Each subject received one tablet of Ambien® 10 mg after an overnight fast of at least 10 hours and a standardized, high fat breakfast.
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Number analyzed (Participants) | 35 | 35
ng/mL | 123.61 (42.45) | 131.92 (45.02)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Zolpidem Tartrate
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable zolpidem tartrate concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Number analyzed (Participants) | 35 | 35
ng-hr/mL | 518.69 (194.66) | 518.68 (184.35)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]for Zolpidem Tartrate
Description: The area under the zolpidem tartrate plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing (hour 0), then 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 4, 5, 6, 8, 10, and 12 hours after dose administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Number analyzed (Participants) | 35 | 35
ng-hr/mL | 560.88 (234.32) | 561.96 (230.63)

ADVERSE EVENTS:
Time Frame: 38 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving both interventions. 36 subjects were administered Zolpidem 10 mg Tablets and 37 subjects were administered Ambien® 10 mg Tablets.
Groups:
- Zolpidem Tartrate 10 mg Tablets; Ambien® 10 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either zolpidem tartrate 10 mg or Ambien® 10 mg following an overnight fast and a standardized, high fat breakfast.
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 9/36 | 6/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem Tartrate 10 mg Tablets (N=36) | Ambien® 10 mg Tablets (N=37)
Blurred vision (Nervous system disorders) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Lightheadedness (Nervous system disorders) | 5 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 1 (1)
Shakiness (Nervous system disorders) | 1 (1) | 0 (0)
Unsteadiness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days